CLINICAL TRIAL: NCT00959062
Title: New Approaches to Pediatric Sedation: Adjunctive Clonidine in the Sedation of Mechanically Ventilated Children (NAPS Pilot Trial)
Brief Title: Adjunctive Clonidine in the Sedation of Mechanically Ventilated Children
Acronym: NAPS Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIF09213
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Respiration, Artificial; Critical Illness; Conscious Sedation; Deep Sedation
Keywords: Pilot Study; Randomized Controlled Trial; Critically Ill; Child; Pediatric; Clonidine; Sedation
MeSH Terms: conditions — Respiratory Aspiration; Critical Illness | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clonidine (Experimental)
  Interventions: Drug: clonidine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clonidine — 5 mcg/kg (maximum 200 mcg) enterally every 6 hours
  Arms: clonidine
Drug: placebo — Preparation visually identical to clonidine.
  Arms: placebo

SUMMARY:
Almost all critically ill children who are mechanically ventilated require sedation and analgesia. Providing effective sedation for children in the PICU requires careful balancing of the need for sedation with the adverse effects associated with sedative medications. Clonidine is often used as an adjunctive sedative and analgesic in children but a well designed and adequately powered randomized trial is required to test the effect of clonidine-based sedation. Because there are no large randomized trials of sedation related interventions among critically ill children there are many unknown factors. This pilot trial, focussing on feasibility outcomes will assess the feasibility of, and inform the design of, a larger randomized controlled trial which will focus on clinically important outcomes.

DETAILED DESCRIPTION:
Almost all critically ill children who are mechanically ventilated require sedation and analgesia. Providing effective sedation for children in the PICU requires careful balancing of the need for sedation with the adverse effects associated with sedative medications. Inadequate sedation may result in undue pain and suffering for children, ventilator dysynchrony and may risk removal of life sustaining devices. Excess sedation limits patients' interaction with their parents and care-givers and may result in delayed weaning from mechanical ventilation, prolonged PICU stay and the attendant risks of increased morbidity. Critically ill children may also experience withdrawal when these medications are stopped. Randomized trails in adults have shown that sedation related interventions can improve patients outcomes, but such trials have not been performed in children.

Clonidine is often used as an adjunctive sedative and analgesic in children but a well designed and adequately powered randomized trial is required to test the effect of clonidine-based sedation. Because there are no large randomized trials of sedation related interventions among critically ill children there are many unknown factors.

This pilot trial, focussing on feasibility outcomes will assess the feasibility of, and inform the design of, a larger randomized controlled trial which will focus on clinically important outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged 1 month to 18 years
* mechanically ventilated
* the attending physician expects to require mechanical ventilation for at least 2 more days
* requires sedation in the form of: morphine by continuous infusion or greater than 4 intermittent doses in the previous 24 hours or fentanyl as a continuous infusion AND midazolam or lorazepam by continuous infusion or more than 3 intermittent doses of lorazepam or 6 doses of midazolam in the previous 12 hours
* has enteral access (gastric or jejunal feeding tube)

Exclusion Criteria:

* hemodynamically unstable
* meet the American College of Critical Care Medicine hemodynamic definition of shock
* hypotensive or tachycardic
* bradycardia, hemodynamically significant cardiac disease or chronic use of anti-hypertensive or diuretic medications
* a traumatic brain injury on admission
* chronically (defined as routine administration prior to hospital admission or for greater than 7 days in hospital prior to PICU admission) use benzodiazepines or opioids
* have received greater than two doses of clonidine within the previous 2 days or dexmedetomidine in the past 2 days
* were previously enrolled in this study
* are currently enrolled in a related study
* are known to be pregnant or breastfeeding
* are known to be allergic to clonidine or any other ingredient in the tablets or suspension
* are being considered for organ procurement
* were chronically (>30 days) ventilated prior to PICU admission
* are currently receiving, or are expected to initiate the ketogenic diet
* are receiving cyclosporine or methylphenidate

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of screening procedures. | 90 days
Protocol adherence. | 90 days
Enrollment rate. | 90 days
Timeliness of drug administration. | 90 days

SECONDARY OUTCOMES:
Sedation and analgesia requirements. | 90 days
Opioid and/or benzodiazepine withdrawal symptoms. | 90 days
Adverse effects. | 90 days
Duration of hospital stay. | 90 days
Ventilator-free days (number of days alive and breathing unaided within the first 28 days after intubation). | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Duffett, Principal Investigator — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - McMaster Children's Hospital/Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario

REFERENCES:
- [Result] Duffett M, Choong K, Foster J, Cheng J, Meade MO, Menon K, Cook DJ. Clonidine in the sedation of mechanically ventilated children: a pilot randomized trial. J Crit Care. 2014 Oct;29(5):758-63. doi: 10.1016/j.jcrc.2014.05.029. Epub 2014 Jun 11. PMID 25015006